CLINICAL TRIAL: NCT04871438
Title: Flash CONtinous Glucose Monitoring in TRansition to Outpatient: Libre for Type 2 Diabetes Mellitus (CONTROL-DM)
Acronym: CONTROL-DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woodlands Health Campus (Other Government)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DSRB 2020/01468
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Flash continuous glucose monitoring; Transitional care; FreeStyle Libre

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FGM (Experimental): Flash glucose monitoring at weeks 0-2, weeks 6-8 post-discharge
  Interventions: Device: Flash glucose monitoring
- SMBG (No Intervention): Self-monitoring of blood glucose at least 4 times a day, 3 days a week

INTERVENTIONS:
Device: Flash glucose monitoring — Group A will use FreeStyle Libre for two weeks of FGM-based titration of medications at two time-points: 1) At recruitment and 2) At 6 weeks. Outside of these time points, they will use SMBG (standard care) for monitoring of blood glucose.
  Other Names: Abbott FreeStyle Libre
  Arms: FGM

SUMMARY:
This is a pilot study of the use of flash glucose monitoring (FGM) to assess glycemic control, behavioural, quality of life benefits and manpower utilization in poorly controlled T2DM patients on insulin in the transitional care period after discharge from hospital.

DETAILED DESCRIPTION:
Background:

Hospitalization often provides an opportunity to optimise the care of patients with diabetes, however, there could be destabilisation of dietary habits and diabetes therapy during admission. During transition from hospital to home, diabetes treatment may be intensified to control hyperglycemia, such as starting insulin therapy, or, de-escalated, due to risks of hypoglycaemia secondary to variable oral intake and physical activity levels peri-hospitalization.

Achieving optimal glycemic control necessitates frequent blood glucose monitoring. However, patients may perceive repeated self-monitoring of blood glucose (SMBG) as inconvenient, intrusive and laborious as it requires pricking their fingers multiple times, resulting in reduced compliance and poorer glycemic outcomes. Ambulatory flash glucose monitoring (FGM) may overcome this and facilitate more rapid achievement of euglycemia due to the benefit of immediate feedback of glucose levels with changes in diet, medication and activity.

As the transitional care period is a period of stress for patients and an opportunity to encourage behavioural change, we propose that the use of intermittent short term FGM in the first two weeks post discharge, and for another two weeks at a 6-week interval may promote behavioural change resulting in improvements in glycemic control.

Objectives:

1. To explore the use of FGM in patients with T2DM with baseline HbA1c >9% and requiring insulin who at risk of hypoglycemia or hyperglycemia, in facilitating the transition care from inpatient to the ambulatory setting.
2. This pilot study is exploratory to determine the logistics and feasibility of the protocol, and to collect preliminary information that will lead to a larger grant application for a larger clinical trial in the future.

Hypotheses:

1. FGM use in patients with T2DM with baseline HbA1c >9% and requiring insulin would facilitate the transition of care from inpatient to the ambulatory setting, resulting in improved glycemic control, as measured by HbA1c at 12 weeks.
2. FGM use in the transitional care period would lead to improved time in range (TIR), reduced time in hypoglycaemia and hyperglycaemia, reduced readmission rates for hypo or hyperglycaemia, improved quality of life, reduced loss to follow-up and encourage individual lifestyle modification, without a significant increase in costs and manpower utilization.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-80 inclusive
* HbA1c>9% on insulin
* Requiring inpatient adjustment of DM medication if meets any of the following:
* A) Hypoglycemia (defined as glucose < 4 mmol/l occurring 2 or more times at least 3 hours apart in the last 72 hours or any glucose <2.5 mmol/l in the last 24 hours)
* B) Hyperglycemia (defined as glucose > 14 mmol/l occurring 2 or more times in the last 36 hours, or any glucose > 24 mmol/l in the last 24 hours)
* Desire to lower HbA1c to a target of 7%
* Willing to wear FGM device
* Willing and able to use FreeStyle Librelink app on personal device
* Willing to avoid use of ascorbic acid throughout the study
* Willing to perform SMBG (by history) of an average of at least 4 times a day, 3 days a week

Exclusion Criteria:

* T1DM
* Pregnant or planning pregnancy during duration of study
* Unable to use or unwilling to comply with study requirements
* Use of personal FGM within 3 months of screening or plan to use personal FGM during the course of the study
* On ascorbic acid
* Extensive skin changes that preclude wearing the sensor on normal skin (e.g. extensive psoriasis, extensive eczema, recent burns or severe sunburn, extensive tattoos, dermatitis herpetiformis)
* Known allergy to medical-grade adhesives
* Renal insufficiency (eGFR<30)
* Pancreatic insufficiency or history of pancreatitis
* Patients on any structured weight reduction interventions such as prescription weight loss medications, bariatric surgery, or protein sparing modified fast during the course of the study.
* Current or anticipated short term uses of glucocorticoids (oral, injectable, or intravenous. Long-term stable glucocorticoid doses are allowed, such as for treatment of rheumatoid arthritis or Addison's disease.
* Any medical condition that would make it inappropriate to target an HbA1c of <7%
* Currently abusing illicit drugs, alcohol or prescription drugs
* Any condition per investigator assessment, that could impact reliability of the HbA1c measurement, such as but not limited to hemoglobinopathy, haemolytic anaemia, chronic liver disease, chronic GI blood loss, recent red blood cell transfusion or erythropoietin administration within 3 months prior to screening
* Current participation in another investigational study (must have completed any prior studies at least 30 days prior to being enrolled in this study)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 weeks, 12 weeks
  Assess change in glycaemic control between groups

SECONDARY OUTCOMES:
% Time in range, % Time below range, % Time above range | 12 weeks
  Glucose in-range defined as 3.9-10.0mmol/l, below range = glucose <3.9mmol/l, above range = glucose >10.0mmol/l
Glycaemic variability | 12 weeks
  Defined by SD and CV
Severe hypoglycemia events | 12 weeks
  Defined by number of hypoglycemic events requiring 3rd party to rescue
Resource utilization | 12 weeks
  Defined as time used for telehealth and clinic consults
Number of re-admissions for dysglycemia or device-related complications | 12 weeks
  Within duration of study
Diabetes Distress Scale (DDS) | 12 weeks
  This 17-item scale lists potential problem areas that people with diabetes may experience, and can denote the degree to which they are or are not affected. Min-Max score of 1-6, where higher score indicates more distress.
Audit of Diabetes-Dependent Quality-of-Life Questionnaire (ADDQoL) | 12 weeks
  This questionnaire assesses the impact of diabetes on 19 life domains including physical functioning, symptoms, psychological well-being, social well-being, role activities and personal constructs, and allows them to indicate the importance of these domains to their quality of life. Average weighted impact score Min to Max -9 to +3, where a lower score indicates poorer quality of life.
Glucose Monitoring Satisfaction Score (GMSS) | 12 weeks
  This 15-item scale evaluates patient satisfaction with their glucose monitoring device and its impact on their quality of life including 4 sub-sections on openness, emotional burden, behavioural burden and worthwhileness. Min-max score of 1-5, where a higher score indicates greater satisfaction.

OTHER OUTCOMES:
Mean glucose | 12 weeks
  Mean glucose
Dietary intake | 12 weeks
  measured in kcal/day
Exercise duration | 12 weeks
  measured in minutes/week

CONTACTS AND LOCATIONS:
Overall Officials: Caroline WS Hoong, Principal Investigator — Woodlands Health Campus
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirschman KB, Bixby MB. Transitions in Care from the Hospital to Home for Patients With Diabetes. Diabetes Spectr. 2014 Aug;27(3):192-5. doi: 10.2337/diaspect.27.3.192. PMID 26246779
- [Background] Rushakoff RJ, Sullivan MM, MacMaster HW, Shah AD, Rajkomar A, Glidden DV, Kohn MA. Association Between a Virtual Glucose Management Service and Glycemic Control in Hospitalized Adult Patients: An Observational Study. Ann Intern Med. 2017 May 2;166(9):621-627. doi: 10.7326/M16-1413. Epub 2017 Mar 28. PMID 28346946
- [Background] Levitt DL, Silver KD, Spanakis EK. Inpatient Continuous Glucose Monitoring and Glycemic Outcomes. J Diabetes Sci Technol. 2017 Sep;11(5):1028-1035. doi: 10.1177/1932296817698499. Epub 2017 Mar 14. PMID 28290224